CLINICAL TRIAL: NCT05784532
Title: Sternal Fixation With STERN FIX After Medial Sternotomy
Status: Withdrawn | Type: Observational
Why Stopped: Participating sites could not perform recruitment due to administrative obstacles that could not be addressed. Sponsor decided in agreement with sites to withdraw the study.
Sponsor: NEOS Surgery (Industry)
Collaborators: Anagram-ESIC (Unknown)
Responsible Party: Sponsor
Other Study IDs: NEO-SC1-2022-01
Record Dates: First submitted 2023-02-20; First posted 2023-03-27 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Sternotomy
Keywords: Rigid Fixation; Sternal Closure; STERN FIX

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- STERN FIX: Patients undergoing cardiothoracic surgery through median sternotomy, once the main intervention is finished, will have their sternum closed using the sternal stabilization system STERN FIX in combination with wires according to the STERN FIX instructions for use.
  Interventions: Device: STERN FIX

INTERVENTIONS:
Device: STERN FIX — Sternotomy closure with STERN FIX and supplemented with wires
  Other Names: Sternal stabilization system

SUMMARY:
The goal of this single arm observational registry is to evaluate the safety and performance of the STERN FIX device in normal conditions of use, in patients treated with medial sternotomy according to the instructions for use.

The main goal of this registry is to evaluate the sternal stability in patients who had their sternum fixed with the STERN FIX system.

Participants will have their sternotomy closed with the STERN FIX device at the end of their cardiothoracic surgery and will be followed up as per standard of care. At discharge and at the 1 month FU visit the sternal stability will be assessed using the sternal instability scale (SIS).

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years old patient
* Patient undergoing surgery requiring medial sternotomy
* Patient able and willing to provide informed consent to participate in the registry and/or who have provided written consent to have their clinical data added to the registry

Exclusion Criteria:

* Patients that are still growing.
* Patients with Sternal anomalies preventing the use of the STERN FIX Sternal Stabilization System, such as bone tumors located in the implant region.
* Patient with conditions previous to surgery that may impact healing, including bone blood supply limitations, insufficient quantity or quality of bone, or other severe structural bone damage.
* Patients with suspected or known allergies or intolerances to the implant material.
* Patients with severe osteoporosis or other degenerative bone diseases.
* Any patient unwilling to, or incapable of, following postoperative care instructions.
* Patients with any other medical or surgical process that may compromise or limit the adequate functionality of the implant.
* Pregnant patients or planning to become pregnant during the 2 months following surgery.
* Patients with life expectancy lower than 2 months.
* Patients who are or have been participating in an interventionist trial during the last 4 weeks

Intraoperative exclusion criteria

* Latent or active infection, or inflammation in the operating area.
* Signs of infection on the surgical site.
* Parasternal sternotomy.
* When the STERN FIX Sternal Stabilization System cannot ensure sufficient fixation.
* When a STERN FIX Sternal Stabilization System device cannot be placed properly in any intercostal space.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All those patients that have or will undergo medial sternotomy during the registry period will be considered for inclusion. They will be informed about it, and if they consent for their data to be used in the registry, their eligibility will be assessed. If a patient does not comply with all IFUs indications, they will not be included in the registry
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Sternal stability | One month postoperatively
  The primary outcome for this registry will be the sternal stability assessed with the sternal instability scale (SIS). The SIS is a scale ranging from 0 to 3 with the following descriptors:
  * 0. Clinically stable sternum (no detectable motion) - normal
  * 1. Minimally separated sternum (slight increase in motion upon special testing* - upper limbs, trunk)
  * 2. Partially separated sternum - regional (moderate increase in motion upon special testing*)
  * 3. Completely separated sternum - entire length (marked increase in motion upon special testing*)

SECONDARY OUTCOMES:
Prevalence and type of AE and SAE | Through study completion, an average of 6 months
  All adverse events occurring during the study period related to the sternotomy must be recorded. The AE that should be recorded, include:
  * Any device complication (wire o STERN FIX fracture, rotation, migration, …)
  * Surgical complications: any injury caused by the devices or instruments.
  * Tissue reactions to implant materials.
  * Damage to the tissues surrounding the devices.
  * Osseous complications (fractures, sternal dehiscence, malunion, nonunion, instability, necrosis, calcification, decrease in bone density….).
  * Postoperative hematoma/ bleeding.
  * Infectious complications (superficial wound infections, mediastinitis, abscess …).
  * Increased fibrous tissue, keloid or seroma formation in the sternotomy area.
  * Any other AE that the investigator considers relevant for the registry.
Prevalence of device deficiencies. | Through study completion, an average of 6 months
  Adverse event related to the use of an investigational medical device. This includes adverse events resulting from insufficient or inadequate instructions for use, deployment, implantation, installation, or operation, or any malfunction and events resulting from use error or from intentional misuse of the investigational medical device.
Sternal closure time | Surgery
  Time elapsed from the measurement of the intercostal spaces to the closure of the last intercostal space.
Easiness of implantation of the device (Likert) | Immediately after surgery
  The easiness score assessed by the surgeon about the usage of the medical device will be registered according to the Likert scale (1-5) with the following descriptors:
  * 5. Very easy
  * 4. Easy
  * 3. Neither easy or difficult
  * 2. Difficult
  * 1. Very difficult
Easiness of implantation of the device (assistance) | Immediately after surgery
  The surgeon will indicate whether they requested external assistance during the implantation of the device
Surgeon satisfaction for the use of the device | Immediately after surgery
  The surgeon general satisfaction with the sternotomy closure using STERN FIX will be assessed in comparison with the usual wire closure using the Likert scale (1-5) with the following descriptors:
  * 5. Very satisfied
  * 4. Satisfied
  * 3. Neither satisfied or dissatisfied
  * 2. Dissatisfied
  * 1. Very dissatisfied

OTHER OUTCOMES:
Performance of the device in high-risk patients (Stability) | One month postoperatively
  The performance of the device (stability) in high-risk patients will be assessed in a sub-analysis.
  Patients considered of high-risk should comply at least one of the following criteria:
  * Pre-operative criteria: diabetes mellitus, COPD, obesity (BMI ≥30kg/m2), renal failure, chronic usage of steroids, immunosuppression, previous sternotomy, osteoporosis.
  * Intra-operative criteria: BIMA, cardiopulmonary bypass lasting more than 2 hours.
  The sternal stability assessed with the sternal instability scale (SIS). The SIS is a scale ranging from 0 to 3 with the following descriptors:
  * 0 Clinically stable sternum (no detectable motion) - normal
  * 1 Minimally separated sternum (slight increase in motion upon special testing* - upper limbs, trunk)
  * 2 Partially separated sternum - regional (moderate increase in motion upon special testing*)
  * 3 Completely separated sternum - entire length (marked increase in motion upon special testing*)
Safety of the device in high-risk patients (AE and SAE prevalence) | Through study completion, an average of 6 months
  The safety of the device (prevalence and type of AE and SAE) in high-risk patients will be assessed in a sub-analysis.
  All adverse events occurring during the study period related to the sternotomy must be recorded. The AE that should be recorded, include:
  * Any device complication (wire o STERN FIX fracture, rotation, migration, …)
  * Surgical complications: any injury caused by the devices or instruments.
  * Tissue reactions to implant materials.
  * Damage to the tissues surrounding the devices.
  * Osseous complications (fractures, sternal dehiscence, malunion, nonunion, instability, necrosis, calcification, decrease in bone density….).
  * Postoperative hematoma/ bleeding.
  * Infectious complications (superficial wound infections, mediastinitis, abscess …).
  * Increased fibrous tissue, keloid or seroma formation in the sternotomy area.
  * Any other AE that the investigator considers relevant for the registry.

CONTACTS AND LOCATIONS:
Locations (1):
- New York-Presbyterian Hospital, Ney York, New York, United States

IPD SHARING:
Plan to Share IPD: No